CLINICAL TRIAL: NCT01605344
Title: A Prospective, Randomized, Crossover Evaluation of the Effect of Atorvastatin on the Pharmacokinetics of Irinotecan in Colorectal Cancer Patients Receiving FOLFIRI
Brief Title: Crossover Evaluation of Effect of Atorvastatin on PK of Irinotecan in CRC Patients Receiving FOLFIRI
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was withdrawn due to lack of patient enrollment.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LCCC 1127
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Advanced Adenocarcinoma of the Colon or Rectum
Keywords: Advanced colon cancer; Advanced rectal cancer; Metastatic colon cancer; Metastatic rectal cancer; Lipitor; Atorvastatin; FOLFIRI
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — IFL protocol; Fluorouracil; Leucovorin; Irinotecan; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): ARM A subjects will receive atorvastatin 20 mg orally once daily given for two weeks prior to FOLFIRI. The last dose of atorvastatin will be taken day 1 of FOLFIRI. ARM A will then receive no statin for the next 2 weeks. Patients will receive FOLFIRI infusion on day 1 and day 15. Blood samples will be collected at baseline and periodically through 24 hours on day 1 and 15 of FOLFIRI.
  Interventions: Drug: FOLFIRI.; Drug: Atorvastatin
- Arm B (Experimental): ARM B subjects will receive no atorvastatin prior to day 1 of FOLFIRI. ARM B subjects will receive atorvastatin 20 mg orally once daily for two weeks prior to day 15 of FOLFIRI. The last dose of atorvastatin will be taken day 15 of FOLFIRI. Patients will receive FOLFIRI infusion on day 1 and day 15. Blood samples will be collected at baseline and periodically through 24 hours on day 1 and 15 of FOLFIRI.
  Interventions: Drug: FOLFIRI.; Drug: Atorvastatin

INTERVENTIONS:
Drug: FOLFIRI. — All patients will receive FOLFIRI infusion on day 1 and day 15.
  Other Names: 5-fluorouracil + leucovorin + irinotecan
Drug: Atorvastatin — A subjects will receive atorvastatin 20 mg orally once daily given for two weeks starting on Day -14 during PERIOD ONE. ARM A will then receive no statin during PERIOD TWO. ARM B subjects will receive no atorvastatin during PERIOD ONE. ARM B subjects will receive atorvastatin 20 mg orally once daily for two weeks during PERIOD TWO (starting on Day 2). One cycle = 28 days.
  Other Names: Lipitor

SUMMARY:
The purpose of this study is to evaluate the effect of atorvastatin on the pharmacokinetic profile of irinotecan and SN-38. To further evaluate the safety of atorvastatin in combination with FOLFIRI. To further evaluate the safety and of irinotecan in combination with atorvastatin.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized, crossover study to address the pharmacokinetic effects of atorvastatin on irinotecan metabolism in patients receiving their first cycle of FOLFIRI (5-fluorouracil + leucovorin + irinotecan).

Each cycle of FOLFIRI is defined as 28 days, with a dose of FOLFIRI administered on day 1 and day 15. Patients will be recruited from the UNC Lineberger Cancer Center, referred by their primary oncologist for the treatment of metastatic colorectal cancer (mCRC). After obtaining informed consent, the patient will be randomized to either ARM A or ARM B.

Blood samples will be collected on day 1 and 15 of FOLFIRI prior to treatment with irinotecan (baseline), immediately following the end of the irinotecan infusion, and at 0.5, 1, 1.5, 2, 4, 6, and 24 hours following the end of the irinotecan infusion.

ARM A subjects will receive atorvastatin 20 mg orally once daily given for two weeks starting on Day -14 during PERIOD ONE. ARM A will then receive no statin during PERIOD TWO. Patients will receive FOLFIRI infusion on day 1 and day 15. Blood samples will be collected at baseline and periodically through 24 hours.

ARM B subjects will receive no atorvastatin during PERIOD ONE. ARM B subjects will receive atorvastatin 20 mg orally once daily for two weeks during PERIOD TWO (starting on Day 2). Patients will receive FOLFIRI infusion on day 1 and day 15. Blood samples will be collected at baseline and periodically through 24 hours.

DNA extraction and genetic analysis of UGT1A1 polymorphisms will be performed in collaboration with Dr. Federico Innocenti and those patients homozygous for the UGT1A1*28 allele will be excluded due to their altered irinotecan metabolism.

Patients will be followed until Day 1 of Cycle 2 of FOLFIRI. Patients removed from study for unacceptable adverse events will be followed until resolution or stabilization of the event(s).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age (no upper age limit)
2. Histological or cytological documentation of adenocarcinoma of the colon or rectum, and patient scheduled to begin FOLFIRI for treatment of their metastatic disease
3. Patients taking statins at the time of enrollment are permitted. Patients taking statins (or one of the prohibited drugs, see section 4.2.27 and section 12.1) must agree to a 2 week washout prior to treatment with atorvastatin (see Schema) and section 5.2
4. Life expectancy of at least 3 months
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
6. Adequate bone marrow, renal, and hepatic function, as evidenced by the following within 7 days of treatment initiation with atorvastatin (or nothing, if enrolled into Arm B): absolute neutrophil count (ANC) ≥1,500/mm3 platelets ≥100,000/mm3 hemoglobin ≥9.0 g/dL serum creatinine ≤1.5 x upper limit of normal (ULN) AST and ALT ≤ 3 x ULN Total bilirubin ≤ 1.5 x ULN Alkaline phosphatase ≤2.5 x ULN Amylase and lipase ≤1.5 x ULN INR/PTT ≤1.5 x ULN CPK ≤ ULN
7. Women of childbearing potential and male subjects must agree to use adequate contraception for the duration of study participation. Adequate contraception is defined as any medically recommended method (or combination of methods) as per standard of care.
8. Medical oncologist agrees that two week window is appropriate/safe prior to start of FOLFIRI for trial candidate.
9. The subject is capable of understanding and complying with parameters as outlined in the protocol
10. Signed, IRB-approved written informed consent

Exclusion Criteria:

1. Any prior allergies to statin therapy or adverse events that precluded further use, including but not limited to myopathy, rhabdomyolysis, etc. Patients who had to change from atorvastatin to another statin for safety or efficacy reasons will also be excluded.
2. Prior treatment with FOLFIRI or single agent irinotecan is prohibited within six weeks of enrollment. All prior toxicity from previous irinotecan administration must be resolved prior to enrollment. No more than 2 prior therapeutic regimens for metastatic disease are allowed.
3. Patients will not be allowed to receive bevacizumab or EGFR inhibitors (cetuximab or panitumumab) for the duration of the study (1 cycle).
4. Patients with baseline LDL ≤ 100 mg/dL who are not currently treated with statins
5. Patients homozygous for the UGT1A1*28 allele, and patients of Asian descent homozygous or heterozygous for the UGT1A1*6 allele will be excluded due to their altered irinotecan metabolism
6. Pregnant or breastfeeding patients. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of atorvastatin and FOLFIRI treatment, and a negative result must be documented before start of treatment with atorvastatin or FOLFIRI (whichever is received first by patient).
7. Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated ≥2 weeks prior to enrollment, may be continued.
8. History of Gilbert's syndrome
9. Pernicious anemia or other anemias due to Vitamin B12 deficiency (due to potential masking of deficiency by leucovorin)
10. Known Dihydropyrimidine dehydrogenase (DPD) deficiency
11. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of Day 1 of treatment with FOLFIRI
12. Any patients with a history of stroke or TIA within 6 months prior to study enrollment
13. Active cardiac disease including any of the following: Congestive heart failure (New York Heart Association [NYHA]) ≥Class 2 (see Appendix C) Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months). Myocardial infarction less than 6 months before start of Day 1 of FOLFIRI Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
14. Ongoing infection > Grade 2 according to NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v. 4.0)
15. Known history of human immunodeficiency virus (HIV) infection
16. Presence of acute or chronic liver disease, renal disease or pancreatitis
17. Known history of chronic hepatitis B or C
18. Symptomatic metastatic brain or meningeal tumors unless the patient is >6 months from definitive therapy, has a negative imaging study within 4 weeks of FOLFIRI initiation, and is clinically stable with respect to the tumor at the time of study entry. Also, the patient must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable provided that the dose is s4.2.2table for one month prior to D1 of treatment under this study)
19. History of organ allograft
20. Non-healing wound, ulcer, or bone fracture
21. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation
22. Inability to swallow oral medications
23. Evidence or history of bleeding diathesis. Any hemorrhage or bleeding event > Grade 4 within 4 weeks of start of FOLFIRI
24. Patients with diarrhea CTCAE v4 grade ≥2
25. Any malabsorption condition
26. Unresolved toxicity higher than CTCAE v. 4.0 Grade 1 attributed to any prior therapy/procedure excluding alopecia and oxaliplatin-induced neurotoxicity (which must be ≤Grade 2)
27. Patients unable or unwilling to discontinue (and substitute if necessary) use of prohibited drugs, juices and herbal supplements for at least 2 weeks prior to atorvastatin initiation (see Appendix A for list of prohibited drugs, juices and herbal supplements)
28. Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
29. Unwilling to provide consent for genetic studies of whole blood or plasma specimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of irinotecan. | Blood samples will be collected on day 1 and 15 of FOLFIRI prior to treatment with irinotecan (baseline), immediately following the end of the irinotecan infusion, and at 0.5, 1, 1.5, 2, 4, 6, and 24 hours following the end of the irinotecan infusion.
  At the end of the screening period, eligible patients will be randomly assigned in a 1:1 ratio to receive atorvastatin prior to Day 1 of FOLFIRI (ARM A) or atorvastatin prior to Day 15 FOLFIRI (ARM B). Patients in ARM A must start atorvastatin within 28 days of randomization and patients in ARM B should receive FOLFIRI within 28 days of randomization; if not, the Investigator must be notified.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of SN-38. | Blood samples will be collected on day 1 and 15 of FOLFIRI prior to treatment with irinotecan (baseline), immediately following the end of the irinotecan infusion, and at 0.5, 1, 1.5, 2, 4, 6, and 24 hours following the end of the irinotecan infusion.
  At the end of the screening period, eligible patients will be randomly assigned in a 1:1 ratio to receive atorvastatin prior to Day 1 of FOLFIRI (ARM A) or atorvastatin prior to Day 15 FOLFIRI (ARM B). Patients in ARM A must start atorvastatin within 28 days of randomization and patients in ARM B should receive FOLFIRI within 28 days of randomization; if not, the Investigator must be notified.

CONTACTS AND LOCATIONS:
Overall Officials: Autumn McRee, MD, Principal Investigator — University of North Carolina at Chapel Hill Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina at Chapel Hill Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Website for UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org